CLINICAL TRIAL: NCT02283476
Title: The Comparative Study on Rh-Endostatin (Endostar®) Continuous Intravenous Infusion and Routine i.v in Combination With GP Regimens for Phase III B/IV Squamous Cell Lung Cancer and Biological Markers Exploration.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM-ED-1302
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Lung Cancer
Keywords: efficacy and safety
MeSH Terms: conditions — Lung Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endostar continuous intravenous infusion (Experimental): Endostar continuous intravenous infusion in combination with Gemcitabine and Cisplatin
  Interventions: Drug: Endostar continuous intravenous infusion; Drug: Gemcitabine; Drug: Cisplatin
- Endostar routine intravenous infusion (Active Comparator): Endostar routine intravenous infusion in combination with Gemcitabine and Cisplatin
  Interventions: Drug: Endostar routine intravenous infusion; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Endostar continuous intravenous infusion — Endostar,7.5mg/m2, continuous intravenous infusion for 14 days each cycle, 21 days as one cycle, 4 cycles in total.
  Arms: Endostar continuous intravenous infusion
Drug: Endostar routine intravenous infusion — Endostar,7.5mg/m2, routine intravenous infusion 3-4 hours daily each cycle,21 days as one cycle, 4 cycles in total
  Arms: Endostar routine intravenous infusion
Drug: Gemcitabine — Gemcitabine,1000-1250mg/m2,i.v d1,d8 in each cycle,21 days as one cycle, 4 cycles in total
Drug: Cisplatin — Cisplatin,75mg/m2,i.v d1 or d1-3 in each cycle,21 days as one cycle, 4 cycles in total

SUMMARY:
Endostar is a anti-angiogenesis product and has been launched in China . The efficacy and safety have been defined. However, the compliance is unsatisfactory since routine i.v of Endostar is needed for 3 to 4 hours daily during one cycle of 14 days. The continuous intravenous infusion by using venous pump can improve the compliance.The comparative study in efficacy and safety has not been done concerning continuous and routine i.v.In addition, what patient can be benefited from Endostar have not been investigated. The biological markers, such as circulating endothelial cells，CECs, will be explored in the study.

ELIGIBILITY:
Inclusion Criteria:

1. primary lung squamous carcinoma confirmed by cytology and histology, excluding sputum examination.
2. phase IIIB /IV based on IASLC 2009 TNM criteria.
3. at least one measurable tumor based on RECIST 1.1 ( longest diameter: ≥20 mm by CT scan or 10 mm by spiral CT )
4. male or female, age≥18 or ≤75 years old
5. ECOG PS: 0 or 1
6. estimated time of survival: ≥ 3 months
7. suitable hematologic function: ANC≥2×109/L, PLC≥100×109/L and Hb≥9 g/dL
8. suitable liver function: Total bilirubin≤normal ULN, AST and ALT≤2.5×normal ULN, ALP≤5×normal ULN.
9. suitable renal function: Cr≤normal ULN,or Ccr≥60 ml/min
10. EKG normal
11. without no healing wound
12. no history of anti-cancer therapy, or adjuvant/neo-adjuvant chemotherapy for non-metastatic tumor finished for more than 6 months before enrolment.
13. for the female subject with productive ability, urine pregnancy test must be done and is negative within 7 days before enrolment.
14. no history of serious allergic to biologic agents, especially E.Coli products
15. the authorized ICF must be signed

Exclusion Criteria:

1. Woman in pregnancy and breast-feeding, or having productive ability without contraception.
2. Having the serious acute infection uncontrolled or purulent/chronic infection with unhealed wound.
3. Having the serious heart disease, including congestive heart failure, uncontrolled high-risk arrhythmia, unstable angina, myocardial infarction, valvular disease, and refractory hypertension.
4. Having uncontrolled nervous or mental disease with low compliance and reluctance to description of response; uncontrolled primary brain tumor or other metastatic brain cancer with obvious intracranial hypertension or mental symptoms.
5. Having the tendency of bleeding, such as FIB<2G/L
6. Being receiving adjuvant chemotherapy.
7. On other conditions investigator considers, the subject is not fitful to participate the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
objective response rate based on Recist 1.1 edition | 3 months
progress free survival | 18 months

SECONDARY OUTCOMES:
overall survival | 24 months
Quality of life (QoL) Questionnaire | 24 months

OTHER OUTCOMES:
biological marker: CECs | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital, Tianjin, China